CLINICAL TRIAL: NCT05336006
Title: Clinical (BMI & MRI) and Biochemical (Adiponectin, Leptin, TNF-α & IL-6) Effects of High-intensity Aerobic Training With a High Protein Diet in Children With Obesity Following COVID-19 Infection.
Brief Title: Exercise and Diet for Pediatric Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Gopal Nambi, Associate Professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RHPT/020/058
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Pediatric Obesity; COVID-19
Keywords: aerobic training; biochemical; children with obesity; COVID-19; high protein diet
MeSH Terms: conditions — Pediatric Obesity; COVID-19 | interventions — Diet, High-Protein; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity aerobic training with high protein diet - Group A (Experimental): High-intensity aerobic training (HAT) was given at 50 to 70 percent of maximum heart rate. Subsequent to stretching, the subjects were asked to do 30 mins of HAT exercises; consisting of 20 mins on the treadmill and 10 mins on a cycle ergometer at 50 to 70 % of MHR, lastly, 10 mins of cool down was performed.
  Next the participants, in this group A were prescribed with strength training exercises with resistance depending upon each subject's individual muscle assessment.
  In addition to these physical training exercises, this group also received a high protein diet in the range of 1.1 - 1.3 g/kg protein/ ideal body weight/day (>1 g/kg aBW/d), as prescribed by a qualified nutritionist.
  Interventions: Other: High-intensity aerobic training with high protein diet
- Control group - Group B (Placebo Comparator): This group is considered a control group and they were allowed to follow their regular physical activities and dietary pattern.
  Interventions: Other: Control group

INTERVENTIONS:
Other: High-intensity aerobic training with high protein diet — High-intensity aerobic training (HAT) was given at 50 to 70 percent of maximum heart rate. Subsequent to stretching, the subjects were asked to do 30 mins of HAT exercises; consisting of 20 mins on the treadmill and 10 mins on a cycle ergometer at 50 to 70 % of MHR, lastly, 10 mins of cool down was performed.
  Next the participants, in this group A were prescribed with strength training exercises with resistance depending upon each subject's individual muscle assessment.
  In addition to these physical training exercises, this group also received a high protein diet in the range of 1.1 - 1.3 g/kg protein/ ideal body weight/day (>1 g/kg aBW/d), as prescribed by a qualified nutritionist.
  Arms: High-intensity aerobic training with high protein diet - Group A
Other: Control group — This group is considered a control group and they were allowed to follow their regular physical activities and dietary pattern.
  Arms: Control group - Group B

SUMMARY:
The coronavirus disease (COVID-19), is a communicable pandemic disease as stated by the world health organization (WHO), which has been affecting the world since December 2019. COVID-19 infected children develop the signs and symptoms of the disease, which can be exaggerated or life-threatening when associated with comorbidities like; obesity, sickle cell anemia, immune disorders, chromosomal abnormalities, chronic respiratory or cardiac problems, and congenital malformations.3 It is observed that children affected with COVID-19 who are physically inactive or in a sedentary lifestyle may induce and develop obesity. It is a major health concern in this pandemic situation, which can be addressed and treated with the use of appropriate physical training and proper dietary habits.

DETAILED DESCRIPTION:
Children confirmed with COVID-19 infection have some systemic illness, that might lead to children with obesity. They are advised to perform regular physical training and consume a proper diet to prevent and treat negative consequences. Therefore, different obesity management and weight reduction protocols are developed to control and prevent health problems and socio-economic issues associated with obesity. The management of this clinical condition has received very little attention, there is no well-defined exercise protocols or dietary prescription for this special population; therefore, there is a need for an elaborative trial in this field. Hence, the aim of this trial was to investigate and compare the clinical and psychological effects of integrated physical training with a high protein diet versus a low protein diet in community-dwelling COVID-19 infected children with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Positively diagnosed COVID-19 children
* age group of 5 - 12 years
* Body mass index (BMI) between 85th to 99th percentiles

Exclusion Criteria:

* history of physical training,
* taking medications,
* recent surgeries,
* fractures and joint problems in the lower extremity,
* cardiac and respiratory problems,
* neurological issues,
* major psychiatric problems,
* other systemic diseases,
* contraindications for physical training and family with food restrictions

Ages: 5 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | At baseline
  For children, age adjusted BMI percentile (BMI %) was calculated, which is a reliable and valid measurement to measure the stage of obesity.
Body mass index (BMI) | 8 weeks
  For children, age adjusted BMI percentile (BMI %) was calculated, which is a reliable and valid measurement to measure the stage of obesity.
Body mass index (BMI) | 6 months
  For children, age adjusted BMI percentile (BMI %) was calculated, which is a reliable and valid measurement to measure the stage of obesity.

SECONDARY OUTCOMES:
Muscle cross sectional area - CSA | At baseline
  Muscle CSA is measured with Magnetic resonance imaging (MRI) scan, it is an expensive measurement. The CSA of three major muscle such as; half way at arm - biceps, thigh - quadriceps and calf muscles were measured and included for analysis.
Muscle cross sectional area - CSA | 8 weeks
  Muscle CSA is measured with Magnetic resonance imaging (MRI) scan, it is an expensive measurement. The CSA of three major muscle such as; half way at arm - biceps, thigh - quadriceps and calf muscles were measured and included for analysis.
Muscle cross sectional area - CSA | 6 months.
  Muscle CSA is measured with Magnetic resonance imaging (MRI) scan, it is an expensive measurement. The CSA of three major muscle such as; half way at arm - biceps, thigh - quadriceps and calf muscles were measured and included for analysis.
Adiponectin | At baseline
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker Adiponectin levels were measured with ELISA kit
Adiponectin | 8 weeks
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker Adiponectin levels were measured with ELISA kit
Adiponectin | 6 months
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker Adiponectin levels were measured with ELISA kit
Leptin | At baseline
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker Leptin levels were measured with ELISA kit
Leptin | 8 weeks
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker Leptin levels were measured with ELISA kit
Leptin | 6 months
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker Leptin levels were measured with ELISA kit
TNF-α | At baseline
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker TNF-α levels were measured with ELISA kit
TNF-α | 8 weeks
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker TNF-α levels were measured with ELISA kit
TNF-α | 6 months.
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical markers TNF-α levels were measured with ELISA kit
IL-6 | At baseline
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker IL-6 levels were measured with ELISA kit
IL-6 | 8 weeks
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker IL-6 levels were measured with ELISA kit
IL-6 | 6 months.
  Fasting (less than 12 hrs) venous blood samples were collected from all the participants and centrifugation of the specimen was done. Serum and plasma were separated and stored immediately at -800C. Biochemical marker IL-6 levels were measured with ELISA kit

CONTACTS AND LOCATIONS:
Locations (1):
- Gopal Nambi, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
The master data and other study information can be obtained by contacting the principal investigator.